CLINICAL TRIAL: NCT06722157
Title: Randomized, Double-masked, Active-controlled, Multicenter Study to Evaluate Efficacy and Safety of Two Regimens of Intravitreal BI 771716 Against Pegcetacoplan in Participants With Geographic Atrophy Secondary to Age-related Macular Degeneration VERDANT Trial
Brief Title: A Study to Test Whether BI 771716 Helps People With an Advanced Form of Age-related Macular Degeneration (AMD) Called Geographic Atrophy
Acronym: VERDANT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1497-0002; U1111-1308-7923 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Macular Degeneration, Age-related; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — pegcetacoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: BI 771716 (Experimental)
  Interventions: Drug: BI 771716
- Arm B: BI 771716 and Sham comparator (Experimental)
  Interventions: Drug: BI 771716; Drug: Sham comparator to BI 771716
- Arm C: Pegcetacoplan (Active Comparator)
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: BI 771716 — BI 771716
  Arms: Arm A: BI 771716; Arm B: BI 771716 and Sham comparator
Drug: Pegcetacoplan — Pegcetacoplan
  Other Names: Syfovre ®
  Arms: Arm C: Pegcetacoplan
Drug: Sham comparator to BI 771716 — Sham comparator to BI 771716
  Arms: Arm B: BI 771716 and Sham comparator

SUMMARY:
This study is open to people 50 years or older with an eye condition called geographic atrophy. The purpose of this study is to compare a medicine called BI 771716 with a medicine called pegcetacoplan. BI 771716 is being developed to treat people with geographic atrophy. Pegcetacoplan is a medicine already used to treat people with geographic atrophy.

In this study, participants receive either BI 771716 or pegcetacoplan as injections in the eye.

Participants are in the study for a little longer than a year and visit the study site every 4 weeks. At the visits, the study doctor checks the eyes of the participants. The results are compared between the groups of participants to see whether the treatment works. The study doctor also regularly checks participants' health and takes note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Age at least 50 years old at the time of randomization visit
* Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male or female participants. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of use are provided in the participant information. Male participants must be ready and able to use either a condom or abstinence as contraceptive measures
* Diagnosis of geographic atrophy (GA) secondary to age-related macular degeneration (AMD), where the total GA lesion area must be ≥2.5 square millimetres (mm²) and ≤17.5 mm² as measured by Fundus autofluorescence (FAF)

  * If multiple lesions are present in the study eye, at least 1 lesion must have an area of ≥1.25 mm²
  * Note: Fellow eye is not required to have GA
  * Note: subfoveal GA lesions (defined as GA lesions within 1 micron of the foveal center point) will be allowed to be enrolled until a maximum of approximately 60% of participants with subfoveal GA lesions are enrolled. Participants with subfoveal GA lesions already in screening at the time the cap has been reached may be considered for randomization.
* Fellow eye must have sufficient visual function compared to the study eye, per the investigator's medical judgment in consultation with the patient, to support the patient's daily functioning
* BCVA letter score of ≥24 letters, using the ETDRS chart in the study eye (equivalent to ≥20/320 on the Snellen chart). Note: If both eyes meet eligibility criteria, the eye with the worse visual function per the investigator's medical judgment in consultation with the patient, will be selected as the study eye. If both eyes have similar visual function, the study eye will be selected per the investigator's medical judgment in consultation with the patient
* further inclusion criteria apply

Exclusion criteria

* GA lesions whose area cannot be accurately defined in the study eye
* Exudative neovascular AMD (eAMD) in the study eye

  -- Note: eAMD in the fellow eye is allowed. However, if the fellow eye is to be considered for microperimetry and other analyses (as defined in the trial statistical analysis plan), then eAMD is not allowed in either eye.
* Previously received treatment in the study eye for GA secondary to AMD within 4 months or 5 half-lives prior to baseline, whichever is longer
* Previously received an investigational medication (oral or intravitreal) for GA secondary to AMD within 4 months or 5 half-lives prior to baseline, whichever is longer
* Currently enrolled in another investigational device or drug trial, or 30 days or 5 half-lives, whichever is longer since ending another investigational device or drug trial(s) or receiving other investigational treatment(s). Any previous use of gene therapy or cell therapy is not permitted
* Additional eye disease as follows:

  * Any eye disease in the study eye that could compromise BCVA
  * Uncontrolled glaucoma or ocular hypertension with intraocular pressure >24 millimetre of mercury (mmHg) in study eye
  * History of high myopia >8 diopters in the study eye
  * Anterior segment and vitreous abnormalities that would preclude adequate observation with spectral domain optical coherence tomography in the study eye
  * Ocular conditions at the discretion of the investigator that might interfere with outcome of the trial in the study eye
  * Active intraocular inflammation in the study eye
  * Active infectious conjunctivitis in either eye
* Prior vitrectomy surgery in the study eye
* History of major intraocular surgeries including major corneal surgery. Uneventful cataract surgery, refractive surgery, oculoplastic surgery, strabismus surgery, and other extraocular surgery may be permitted if they have occurred more than 3 months prior to baseline in the study eye
* further exclusion criteria apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Slope of change from baseline in square root transformed geographic atrophy (GA) area as measured by fundus autofluorescence (FAF) in the study eye expressed in millimeter (mm)/year | At Baseline , at Week 56

SECONDARY OUTCOMES:
Change from baseline in square root transformed GA area as measured by FAF in the study eye expressed in mm | At Baseline, at Week 56
Change from baseline in best corrected visual acuity (BCVA) as measured by standardized early trial diabetic retinopathy study (ETDRS) chart in the study eye | At Baseline, at Week 56
Occurrence of BCVA letter loss of ≥15 letters as measured by standardized ETDRS chart in the study eye for at least 2 consecutive visits | Up to Week 56
Occurrence of exudative neovascular age-related macular degeneration (eAMD) in the study eye from first drug administration until Week 56 | Up to Week 56
Occurrence of drug-related adverse events (AE) from first drug administration until Week 56 | Up to Week 56

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Associated Retina Consultants, Gilbert, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Phoenix Retina Associates, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Global Research Management, Glendale, California
  - Retina Associates of Southern California, Huntington Beach, California
  - Retinal Consultants Medical Group, Inc, Modesto, California
  - Eye Research Foundation, Newport Beach, California
  - Retina Consultants of San Diego, Poway, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Bay Area Retina Associates - Walnut Creek, Walnut Creek, California
  - Colorado Retina Associates, Lakewood, Colorado
  - Connecticut Eye Consultants, PC, Danbury, Connecticut
  - Retina Group of New England, PC, Waterford, Connecticut
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - University Retina and Macula Associates, Lemont, Illinois
  - Illinois Retina Associates - Oak Park, Oak Park, Illinois
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Minnesota, Edina, Minnesota
  - Mississippi Retina Associates, Madison, Mississippi
  - University of Missouri Health System, Columbia, Missouri
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Long Island Vitreoretinal Consultants - Westbury, Westbury, New York
  - Verum Research, LLC, Eugene, Oregon
  - Mid Atlantic Retina - Bethlehem, Bethlehem, Pennsylvania
  - Charleston Neuroscience Institute - Charleston, Charleston, South Carolina
  - Tennessee Retina, Nashville, Tennessee
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas-Beaumont-70319, Beaumont, Texas
  - Retina Consultants of Texas-Bellaire-67493, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina Consultants of Texas - Katy, Katy, Texas
  - Red River Research Partners, LLC, Plano, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Texas - Schertz, Schertz, Texas
  - Retina Consultants of Texas-The Woodlands-67575, The Woodlands, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Spokane Eye Clinic, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com